CLINICAL TRIAL: NCT00654836
Title: A Phase II Study of Carboplatin, Nanoparticle Albumin-Bound Paclitaxel (ABI-007) and Avastin as the First Line Therapy in Metastatic Breast Cancer.
Brief Title: Carboplatin, Paclitaxel, and Bevacizumab in Treating Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Shelly Lo, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200027
Record Dates: First submitted 2008-04-08; First posted 2008-04-09 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage III breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Carboplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin, ABI-007 and Bevacizumab (Experimental): Participants will receive combination carboplatin, nanoparticle albumin-bound paclitaxel (ABI-007-Abraxane), and bevacizumab (Avastin)
  Interventions: Biological: bevacizumab; Drug: Carboplatin; Drug: ABI-007

INTERVENTIONS:
Biological: bevacizumab — Participants will receive bevacizumab 15 mg/kg on days 1,22, and 43.
  Other Names: Avastin
Drug: Carboplatin — Participants will receive a standard carboplatin dose according to their area under the plasma drug concentration-time curve (AUC-6) on days 1, 22, and 43.
  Other Names: Paraplatin
Drug: ABI-007 — Participants will receive ABI-007 (Abraxane) 100mg/m2 on days 1,8, 15, 22, 29, 36,43,and 50.
  Other Names: Abraxane

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving carboplatin and paclitaxel together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and paclitaxel together with bevacizumab works in treating patients with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the progression-free survival of patients with locally recurrent or metastatic breast cancer treated with carboplatin, paclitaxel albumin-stabilized nanoparticle formulation, and bevacizumab as first-line therapy.

Secondary

* To determine the response rate in these patients.
* To determine the overall survival of these patients.
* To evaluate the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive carboplatin IV over 1 hour and bevacizumab IV on days 1, 22 and 43. Patients also receive paclitaxel albumin-bound nanoparticle formulation IV over 30 minutes on days 1, 8 ,15, 22, 29, 36, 43, and 50. Treatment continues in the absence of disease progression or unacceptable toxicity.

Formalin-fixed paraffin-embedded archived tumor tissue samples are assessed by immunohistochemistry (IHC) for various biomarkers. Levels of Notch-1, Notch-4, cyclin A, cyclin B, Jagged-1, and DLL4 in tumor-associated endothelial cells are correlated with response in both estrogen- and progesterone-positive and negative tumors, and independently of p53 status.

After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary adenocarcinoma of the breast

  * Locally recurrent or metastatic disease
* Must have HER-2-negative breast cancer or, if HER-2-positive, must be unable to receive trastuzumab (Herceptin®) or have previously received trastuzumab in the past
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm by conventional techniques or as > 10 mm by spiral CT scan.
* No known CNS disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Postmenopausal status not specified
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (unless bone metastasis is present in the absence of liver metastasis)
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent malignancies within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

Exclusion criteria:

* Pre-existing neuropathy ≥ grade 1
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Serious, non-healing wound, ulcer, or bone fracture
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications)
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association class II-IV congestive heart failure
* History of myocardial infarction or unstable angina within the past 6 months
* History of stroke or transient ischemic attack within the past 6 months
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Significant traumatic injury within the past 28 days
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Proteinuria, as demonstrated by either urine protein:creatinine ratio ≥ 1.0 OR urine dipstick for proteinuria ≥ 2+

  * Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline must demonstrate 24-hour urine protein ≤ 1g
* History of allergy or hypersensitivity to paclitaxel albumin-stabilized nanoparticle formulation, paclitaxel, bevacizumab, carboplatin, albumin, drug product excipients, or chemically similar agents

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No prior chemotherapy for locally recurrent or metastatic disease
* Prior neoadjuvant or adjuvant chemotherapy allowed
* More than 1 week since prior core biopsy or other minor surgical procedure, excluding placement of a vascular access device
* More than 4 weeks since prior and no concurrent major surgical procedure or open biopsy
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 1 year since prior taxane regimen
* No other concurrent investigational agents
* Concurrent anticoagulation allowed, provided the following criteria are met:

  * Stable dose of warfarin or low molecular weight heparin
  * INR within desired range (2-3)
  * No evidence of active bleeding or coagulopathy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent radiotherapy, chemotherapy, immunotherapy, or antitumor hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2012-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Lo, MD, Principal Investigator — Loyola University
Locations (6):
- United States (6):
  - Good Samaritan Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Central Dupage Cancer Center, Winfield, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with metastatic breast cancer were recruited from medical clinics between October 15, 2007 and February 15, 2012
Pre-assignment Details: No enrolled participant was excluded from therapy
Groups:
- Carboplatin, ABI-007 and Bevacizumab: Participants received combination carboplatin, ABI-007 (i.e., a nanoparticle albumin-bound paclitaxel also called Abraxane), and bevacizumab (Avastin). Bevacizumab was administered as 15 mg/kg on days 1, 22, and 43 for patients without hematologic toxicity. For those with hematologic toxicity, bevacizumab was administered as 10mg/kg on day 1 and 15. Similarly, for patients without hematologic toxicity, a standard carboplatin dose according to the participant's area under the plasma drug concentration-time curve (AUC-6) was administered on days 1, 22, and 43. For patients with a hematologic toxicity, carboplatin was only given on day 1. Finally, for those without hematologic toxicity, ABI-007 (Abraxane) 100mg/m2 was administered on days 1,8, 15, 22, 29, 36,43,and 50. Conversely, for patients with hematologic toxicity, Abraxane was administered as 100mg/m2 only on days 1, 8, and 15.
Period: Overall Study
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants are included in the baseline analysis population
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
Number analyzed (Participants) | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.38 [49.25 to 65.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — The ECOG performance status utilizes a five point grading scale from 0 to 5, with higher values indicating worse patient status. (0 = Fully Active, 1 = Restricted in Physically Activity, 2 = Ambulatory and Capable of Self Care, 3 = Limited Self Care, 4 = Completely Disabled, 5 = Dead).
  participants
    ECOG 0 | 22
    ECOG 1 | 7
    ECOG 2 | 1
    Undetermined | 2
Site of Metastatic Disease was Bone [Number; unit: participants]
  Yes | 20
  No | 12
Site of Metastatic Disease was Liver [Number; unit: participants]
  Yes | 14
  No | 18
Site of Metastatic Disease was Loco-regional [Number; unit: participants]
  Yes | 12
  No | 20
Site of Metastatic Disease was Lung [Number; unit: participants]
  Yes | 9
  No | 23
Site of Metastatic Disease was Distant Lymph Nodes [Number; unit: participants]
  Yes | 7
  No | 25
Prior adjuvant therapy was chemotherapy [Number; unit: participants]
  Yes | 17
  No | 15
Prior adjuvant therapy was endocrine therapy [Number; unit: participants]
  Yes | 18
  No | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was measured from treatment initiation to 30 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 30 Months
Population: All enrolled participants are included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
Number analyzed (Participants) | 32
Months | 16 [9.80 to 22.20]

2. Secondary Outcome: Response Rate at End of Treatment
Description: Response to treatment was recorded 30 months following treatment initiation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progressive Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions .
Time Frame: 30 Months
Population: Of the 32 enrolled participants, two participants did not return to the clinic at 30 months for final evaluation of their response to treatment.
Measure: Number; unit: participants
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
Number analyzed (Participants) | 32
participants
  Complete Response (CR) | 2
  Partial Response (PR) | 24
  Stable Disease (SD) | 3
  Progressive Disease (PD) | 1
  Undetermined | 2

3. Secondary Outcome: Overall Survival
Description: Overall survival was measured from treatment initiation to 80 months
Time Frame: 80 Months
Population: All enrolled participants are included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
Number analyzed (Participants) | 32
Months | 21 [13.48 to 28.52]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from all 32 enrolled participants between February 28, 2008 and April 26, 2013
Arm/Group | Carboplatin, ABI-007 and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 24/32
Serious Adverse Events (participants affected / at risk) | 24/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, ABI-007 and Bevacizumab (N=32)
Disease Progression (General disorders) | 24 (24) — All patients died due to natural disease progression.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, ABI-007 and Bevacizumab (N=32)
Abnormal hemoglobin (Blood and lymphatic system disorders) | 15 (15)
Abnormal Leukocytes (Blood and lymphatic system disorders) | 17 (17)
Anorexia (Psychiatric disorders) | 4 (4)
Constipation (Metabolism and nutrition disorders) | 3 (3)
Cough (General disorders) | 2 (2)
Dyspnea (General disorders) | 4 (4)
Hemorrhage of the Nose (Vascular disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 5 (5)
Chest Pain (General disorders) | 4 (4)
Joint Pain (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 2 (2)
Proteinuria (General disorders) | 2 (2)
Thrombosis (General disorders) | 2 (2)
Abnormal Liver Test (AST) (Hepatobiliary disorders) | 2 (5)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to disclose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No